CLINICAL TRIAL: NCT00763165
Title: Periodontal Disease and Cardiovascular Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Colgate Palmolive (Industry)
Responsible Party: William DeVizio/VP - Clinical Research, Colgate Palmolive
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D/06/Dent/99
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2008-10-02 (Estimated); Status verified 2008-09

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Triclosan; Fluorides

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Triclosan; Drug: Fluoride
- B (Placebo Comparator)
  Interventions: Drug: Fluoride

INTERVENTIONS:
Drug: Triclosan — Brush twice daily
  Arms: A
Drug: Fluoride — Brush twice daily
  Arms: A
Drug: Fluoride — Brush twice daily
  Arms: B

SUMMARY:
To access the influence of triclosan dentifrice on the progression of periodontal disease in patients with coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* A minimum of 12 uncrowned teeth other than 3rd molars
* Age 18 to 75 years
* Informed consent

Exclusion Criteria:

* Prosthetic heart valves
* Prosthetic joint replacement
* Previous infective endocarditis
* Requirement for antibiotic cover for dental treatment
* Current treatment with warfarin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2000-11; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Periodontal disease | 3-5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Seymour, BDS, Principal Investigator
Locations (1):
- Discipline of Medicine, Chermside, Australia